CLINICAL TRIAL: NCT03503201
Title: The Value of Chromium Supplementation on Cycles Characteristics of Patients With Polycystic Ovary Syndrome Undergoing Intracytoplasmic Sperm Injection (ICSI).
Brief Title: Effect of Chromium Supplementation on Intracytoplasmatic Sperm Injection (ICSI) Outcomes in Polycystic Ovary Syndrome Ladies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amira S Dieb, Ob/Gyn Lecturer, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1198900
Record Dates: First submitted 2018-04-02; First posted 2018-04-19 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: PCOS
MeSH Terms: interventions — Chromium

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Active Comparator): patients receive chromium supplementation as capsules of 200 micrograms of chromium picolinte (Arab company for pharmaceuticals and medicinal plants) for 2 months before Intracytoplasmic sperm injection cycle
  Interventions: Dietary Supplement: Chromium
- No treatment (No Intervention): patients will not receive chromium supplementation before Intracytoplasmic sperm injection cycle

INTERVENTIONS:
Dietary Supplement: Chromium — chromium supplementation as capsules of 200 micrograms of chromium picolinte (Arab company for pharmaceuticals and medicinal plants) daily for 2 months before ICSI cycle
  Arms: treatment

SUMMARY:
This study is a prospective, double-blind, randomized controlled trial . It included 60 infertile obese patients with polycystic ovary syndrome (PCOS), who are scheduled for intracytoplasmatic sperm injection (ICSI) cycle. The patients will be randomly allocated into two equal groups; Group (A): patients receive chromium supplementation as capsules of 200 micrograms of chromium picolinate (Arab company for pharmaceuticals and medicinal plants), Group (B): no chromium supplementation. Both patients and outcome assessors are blinded to allocated group. All 100 participants underwent similar ICSI cycles. Primary outcome is clinical pregnancy rate per cycle. Secondary outcomes include Body mass index (BMI) and waist/hip ratio (WHR), fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA) index, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), free and total testosterone , Sex Hormone Binding Globulin (SHBG), Free Androgen index (FAI), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2, Days of stimulation , dose of gonadotrophins, number of M II oocytes retrieved, number of grade1and 2 embryos, number of frozen embryos, freeze all cyles, Ovarian Hyperstimulation syndrome (OHSS), Chemical pregnancy rate, clinical pregnancy, twins and abortion.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled trial that is blinded to investigator and outcome assessors. Ethical committee approval is obtained. The study includes infertile obese patients with PCOS diagnosed according to Rotterdam criteria, who are scheduled for ICSI cycle. Patients with body mass index (BMI) 30-35kg/m2 are included.

Women with diabetes, thyroid disorder or other endocrine dysfunctions, uterine abnormalities are excluded.

All patients receive detailed information about the study and informed consent is given by those who accepted to participate in the study. Each patient is subjected to history taking about obstetric history, medical and surgical history and demographic distribution. Full physical examination and 2D transvaginal sonography (TVS) are done on day 2 to 5 of menses to assess antral follicle count (AFC), uterus and adnexa .

All 100 participants are scheduled for ICSI cycles. Randomization is done by withdrawing closed envelopes for each patient into group A and group B . Group (A): patients receive chromium supplementation as capsules of 200 micrograms of chromium picolinate (Arab company for pharmaceuticals and medicinal plants) for 2 months, Group (B): no chromium supplementation.

Antagonist protocol is followed. Gonadotropins as Intramuscular (I.M.) injections of 150-300 (International units) I.U. of highly purified Human Menopausal Gonadotropins daily (Merional, 75 I.U. /vial, IBSA). and Urofollitropin or highly purified human follicle stimulating hormone(Fostimon®, 75 I.U. /vial, IBSA) are give in a ratio of 1:1.The dose is adjusted according to the age, BMI, Antral follicle count (AFC), serum levels of AMH, FSH and ovarian response.

On the sixth day of stimulation , a visit is scheduled to assess the ovarian response ( folliculometry) by TVS. Gonadotrophin releasing hormone antagonist (GnRH antagonist) which is Cetrorelix 0.25mg ( Cetrotide®, 0.25 mg/ vial, Merck Serono, is filled and mixed with diluent from a prefilled syringe with a 20 gauge needle) is given subcutaneously (S.C.) by 27-gauge needle starting from the 6th day of stimulation (fixed antagonist protocol).

Next visits are every other day for follow up using the TVS. The trigger by Human Chorionic Gonadotrophin (HCG)10000 I.U., I.M. ( Pregnyl, Organon) is given when at least 3 follicles reach 18mm in mean diameter or more and E2 level is less than 2500 pg/ml. Ovum retrieval is done 34 hours after HCG injection and embryo transfer using Wallace catheter on day 2 to 3. Luteal support includes natural Progesterone 400 mg 1x2 as rectal suppository, Folic acid 0.5 mg orally once daily, Amoxicillin-Clavulanic Acid 1gm 1x2x7 orally, Progesterone 100 I.M. injections daily for 10 days, Acetylsalicylic Acid (75 mg) orally once daily, metformin 500-1000 mg orally daily .

Quantitative ß- HCG in serum after is done after 14 days of embryo transfer.TVS is performed to detect clinical pregnancy at 6-7 weeks of gestation.

Primary outcome is clinical pregnancy rate per cycle. Secondary outcomes include Body mass index (BMI) and waist/hip ratio (WHR), fasting insulin , fasting plasma glucose, Homeostatic model assessment (HOMA) index, lipid profile ( Triglycerides (TGs), total cholesterol, High density Lipoprotein (HDL), Low density Lipoprotein (LDL), free and total testosterone , Sex Hormone Binding Globulin (SHBG), Free Androgen index (FAI), AntiMullerian Hormone (AMH), Basal Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estradiol (E2, Days of stimulation , dose of gonadotrophins, number of M II oocytes retrieved, number of grade1and 2 embryos, number of frozen embryos, freeze all cyles, Ovarian Hyperstimulation syndrome (OHSS), Chemical pregnancy rate, clinical pregnancy, twins and abortion.

ELIGIBILITY:
Inclusion Criteria:

* infertile obese patients with PCOS diagnosed according to Rotterdam criteria scheduled for ICSI cycle
* patients with BMI 30-35kg/m2

Exclusion Criteria:

* Women with diabetes, thyroid disorder or other endocrine dysfunctions
* Women with uterine abnormalities.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per cycle | 14 weeks
  detection of gestational sac, embryonal pole and fetal pulsations by ultrasonography per cycle

SECONDARY OUTCOMES:
Body mass index | 8 weeks
  The weight in kilograms divided by the squared height in meters
Concentration of fasting insulin | 8 weeks
  Insulin level in serum after fasting for 8 hours measured as mIU/ml
Concentration of free testosterone | 8 weeks
  Free testosterone level in serum measured as ng/dL
Number of days of stimulation with gonadotrophins | 10 weeks
  Days of stimulation with gonadotrophins
Number of ampoules of gonadotrophins | 10 weeks
  total number of ampoules of gonadotrophins
number of MII oocytes retrieved per cycle | 10 weeks
  number of MII oocytes retrieved per cycle
fertilization rate per cycle | 10 weeks
  fertilization rate per cycle
number of embryos | 14 weeks
  number of embryos
grades of embryo quality | 11 weeks
  embryo quality graded as grade I,II,III,IV
chemical pregnancy rate per cycle | 12 weeks
  chemical pregnancy rate per cycle
twins rate per cycle | 14 weeks
  twins rate per cycle
miscarriage rate per cycle | 28 weeks
  miscarriage rate per cycle
Number of frozen embryos | 10 to 11weeks
  Number of frozen embryos
Number of freeze all cycles | 10 to 11weeks
  total number of freeze all cycles
Number of cases with Ovarian Hyperstimulation Syndrome | 12 to 14 weeks
  number of cases diagnosed with Ovarian Hyperstimulation Syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Amira S Dieb, MD, Principal Investigator — KasrAlainiH
Locations (1):
- KasrELAiniH, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No